CLINICAL TRIAL: NCT03924895
Title: A Randomized Phase 3 Study Evaluating Cystectomy With Perioperative Pembrolizumab and Cystectomy With Perioperative Enfortumab Vedotin and Pembrolizumab Versus Cystectomy Alone in Participants Who Are Cisplatin-Ineligible or Decline Cisplatin With Muscle-Invasive Bladder Cancer (KEYNOTE-905/EV-303)
Brief Title: Perioperative Pembrolizumab (MK-3475) Plus Cystectomy or Perioperative Pembrolizumab Plus Enfortumab Vedotin Plus Cystectomy Versus Cystectomy Alone in Participants Who Are Cisplatin-ineligible or Decline Cisplatin With Muscle-invasive Bladder Cancer (MK-3475-905/KEYNOTE-905/EV-303)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Seagen Inc. (Industry); Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-905; MK-3475-905 (Other: MSD); KEYNOTE-905 (Other: MSD); EV-303 (Other: Astellas Protocol Number); PHRR210911-003890 (Other: Philippine Health Research Registry (PHRR)); jRCT2031220686 (Registry Identifier: Japan Registry of Clinical Trials (jRCT)); 2023-504932-16 (Registry Identifier: EU CT); 2031220686 (Other: JRCT); U1111-1290-4057 (Registry Identifier: UTN); 2018-003809-26 (EudraCT Number)
Record Dates: First submitted 2019-04-22; First posted 2019-04-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Urinary Bladder Cancer, Muscle-invasive
Keywords: Muscle-Invasive Bladder Cancer (MIBC); Enfortumab vedotin (EV); Pembrolizumab (MK-3475)
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; Surgical Procedures, Operative; Cystectomy; enfortumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Pembrolizumab + Surgery (Experimental): Participants receive 3 preoperative cycles of pembrolizumab, followed by standard of care surgery, followed by 14 cycles of postoperative pembrolizumab. Each cycle is 21 days.
  Interventions: Drug: Pembrolizumab; Procedure: Surgery (radical cystectomy (RC) plus Pelvic Lymph Node Dissection [PLND])
- Arm B: Surgery alone (Active Comparator): Participants receive standard of care surgery alone.
  Interventions: Procedure: Surgery (radical cystectomy (RC) plus Pelvic Lymph Node Dissection [PLND])
- Arm C: Enfortumab Vedotin + Pembrolizumab + Surgery (Experimental): Participants receive 3 preoperative cycles of enfortumab vedotin + pembrolizumab, followed by standard of care surgery, followed by 6 cycles of postoperative enfortumab vedotin + pembrolizumab, followed by 8 cycles of pembrolizumab alone. Each cycle is 21 days.
  Interventions: Drug: Enfortumab Vedotin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg by intravenous (IV) infusion, given on Day 1 of each 21-day cycle.
  Other Names: KEYTRUDA®; MK-3475
  Arms: Arm A: Pembrolizumab + Surgery
Procedure: Surgery (radical cystectomy (RC) plus Pelvic Lymph Node Dissection [PLND]) — Surgical RC+PLND will be done in accordance with the American Urological Association (AUA)/American Society of Clinical Oncology (ASCO)/American Society for Radiation Oncology (ASTRO)/Society of Urologic Oncology (SUO) guidelines.
  Arms: Arm A: Pembrolizumab + Surgery; Arm B: Surgery alone
Drug: Enfortumab Vedotin — Enfortumab vedotin 1.25 mg/kg by intravenous (IV) infusion, given on Days 1 and 8 of each 21-day cycle.
  Other Names: Padcev; ASG-22CE; ASG-22ME
  Arms: Arm C: Enfortumab Vedotin + Pembrolizumab + Surgery

SUMMARY:
This is a study of perioperative pembrolizumab or enfortumab vedotin in combination with pembrolizumab in participants who are cisplatin-ineligible or decline cisplatin with muscle-invasive bladder cancer (MIBC).

The primary hypothesis is that perioperative pembrolizumab plus radical cystectomy (RC) plus pelvic lymph node dissection (PLND) and perioperative enfortumab vedotin in combination with pembrolizumab plus RC+PLND will achieve superior event-free survival (EFS) compared with RC+PLND alone.

With Amendment 5, outcome measures for programmed cell death ligand 1 (PD-L1) combined positive score (CPS) were removed.

With Amendment 8, the primary outcome measure of pathologic complete response (pCR) rates was changed to a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of urothelial carcinoma/muscle-invasive bladder cancer [MIBC] (cT2-T4aN0M0 or T1-T4aN1M0) with predominant (≥50%) urothelial histology to be confirmed by Blinded Independent Central Review (BICR) (central pathology and/or imaging).
* Clinically nonmetastatic bladder cancer determined by imaging
* Eligible for radical cystectomy (RC) + pelvic lymph node dissection (PLND), and agreement to undergo curative intent standard RC + PLND (including prostatectomy if applicable)
* Ineligible for treatment with cisplatin, as defined by meeting at least one of the following criteria OR be eligible for treatment with cisplatin but decline treatment with cisplatin-based chemotherapy:

  * Impaired renal function with measured or calculated creatinine clearance (CrCl) 30 to 59 mL/min (calculated by Cockcroft-Gault method, Modification of Diet of Renal Disease [MDRD] equations, or measured by 24-hour urine collection)
  * Eastern Cooperative Oncology Group (ECOG) Performance Status 2
  * Common Terminology Criteria for Adverse Events (CTCAE) v.4 Grade ≥2 audiometric hearing loss
  * New York Heart Association (NYHA) Class III heart failure
* Transurethral resection (TUR) of a bladder tumor that is submitted for central pathology assessment and adequate to determine urothelial histology and PD-L1 expression assessment
* ECOG performance status of 0, 1, or 2
* Adequate organ function
* A male participant is eligible to participate if he agrees to use contraception and refrain from donating sperm during the intervention period and for at least 180 days after the last dose of enfortumab vedotin. If the male participants are receiving pembrolizumab only or undergoing surgery only, there are no contraception requirements
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: Not a (woman of childbearing potential) WOCBP or a WOCBP who agrees to use a highly effective contraceptive method or be abstinent from heterosexual intercourse (as their preferred and usual lifestyle) during the intervention period and for at least 120 days after the last dose of pembrolizumab and at least 180 days after the last dose of enfortumab vedotin; whichever comes last. A female participant must agree not to donate eggs during this period as well
* A WOCBP must have a negative highly sensitive pregnancy test within 24 hours before the first dose of study intervention

Exclusion Criteria:

* Known additional nonurothelial malignancy that is progressing or has required active anticancer treatment ≤3 years of study randomization, with certain exceptions
* Has ≥ N2 or metastatic disease (M1) as identified by imaging
* Received any prior systemic treatment, chemoradiation, and/or radiation therapy for muscle-invasive bladder cancer (MIBC) or non-muscle invasive bladder cancer (NMIBC)
* Received prior therapy with an anti-programmed cell death protein 1 (PD-1), anti-programmed death-ligand 1 (PD-L1), or anti-programmed cell death 1 ligand 2 (PD-L2), or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Received prior systemic anticancer therapy including investigational agents within 3 years prior to randomization
* Received any prior radiotherapy to the bladder
* Received a partial cystectomy of the bladder to remove any non-muscle-invasive bladder cancer (NMIBC) or MIBC
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Current participation in or participation in a study of an investigational agent or use of an investigational device within 4 weeks prior to the first dose of study intervention
* Ongoing sensory or motor neuropathy Grade 2 or higher
* Diagnosis of immunodeficiency or receipt of chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug. Physiologic replacement doses of corticosteroids are permitted for participants with adrenal insufficiency.
* Hypersensitivity to monoclonal antibodies (including pembrolizumab) and/or any of their excipients
* Severe hypersensitivity (≥ Grade 3) to enfortumab vedotin or any excipient contained in the drug formulation of enfortumab vedotin
* Active keratitis or corneal ulcerations. Participants with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator
* Active autoimmune disease that has required systemic therapy in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic therapy and is allowed
* Has uncontrolled diabetes
* History of (noninfectious) pneumonitis that required steroids, or current pneumonitis
* Active infection requiring systemic therapy
* Has had an allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) between Arm C and Arm B | Up to approximately 6.75 years
  EFS is defined as the time from randomization to the first occurrence of any of the following events: progression of disease that precludes RC surgery or failure to undergo RC surgery in participants with residual disease (biopsy-proven muscle-invasive bladder cancer [MIBC] will be considered an event regardless of radiographic findings), gross residual disease left behind at the time of surgery, local or distant recurrence as assessed by imaging and/or biopsy, or death due to any cause.

SECONDARY OUTCOMES:
EFS between Arm A and Arm B | Up to approximately 6.75 years
  EFS is defined as the time from randomization to the first occurrence of any of the following events: progression of disease that precludes RC surgery or failure to undergo RC surgery in participants with residual disease (biopsy-proven muscle-invasive bladder cancer [MIBC] will be considered an event regardless of radiographic findings), gross residual disease left behind at the time of surgery, local or distant recurrence as assessed by imaging and/or biopsy, or death due to any cause.
Overall Survival (OS) between Arm C and Arm B | Up to approximately 7.6 years
  OS is defined as the time from randomization to death due to any cause.
OS between Arm A and Arm B | Up to approximately 7.6 years
  OS is defined as the time from randomization to death due to any cause.
Pathologic Complete Response (pCR) Rate between Arm C and Arm B | Up to approximately 5.7 years
  Pathologic complete response rate is defined as the percentage of participants having pCR. pCR is defined as absence of viable tumor (pT0N0) in examined tissue from RC and PLND, as determined centrally.
pCR Rate between Arm A and Arm B | Up to approximately 5.7 years
  Pathologic complete response rate is defined as the percentage of participants having pCR. pCR is defined as absence of viable tumor (pT0N0) in examined tissue from RC and PLND, as determined centrally.
Disease-Free Survival (DFS) | Up to approximately 6.75 years
  DFS is defined as the time from first post-surgery baseline scan until:
  * local or distant recurrence as assessed by imaging and/or biopsy
  * Death due to any cause
Pathologic Downstaging (pDS) Rate between Arm A and Arm B | Up to approximately 5.7 years
  Pathologic downstaging rate is defined as the percentage of participants having pDS. pDS is defined as participants with a tumor classification of <pT2 (includes pT0, pTis, pTa, pT1) and N0 in examined tissue from RC and PLND.
pDS Rate between Arm C and Arm B | Up to approximately 5.7 years
  Pathologic downstaging rate is defined as the percentage of participants having pDS. pDS is defined as participants with a tumor classification of <pT2 (includes pT0, pTis, pTa, pT1) and N0 in examined tissue from RC and PLND.
Number of Participants Experiencing Adverse Events (AEs) | Up to approximately 7.6 years
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Number of Participants Discontinuing Study Drug Due to Adverse Events (AEs) | Up to approximately 1 year
  An AE is defined as any unfavorable and unintended sign, symptom, or disease (new or worsening) temporally associated with the use of study therapy, regardless of whether or not a causal relationship with the study therapy can be determined.
Number of Participants Experiencing Perioperative Complications | Up to approximately 1 year
  The number of participants who experience perioperative complications will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (242):
- United States (39):
  - University of South Alabama, Mitchell Cancer Institute ( Site 1582), Mobile, Alabama
  - CARTI Cancer Center ( Site 1577), Little Rock, Arkansas
  - St. Joseph Heritage Healthcare ( Site 0046), Fullerton, California
  - Scripps MD Anderson ( Site 0010), La Jolla, California
  - Hoag Memorial Hospital Presbyterian ( Site 1595), Newport Beach, California
  - John Wayne Cancer Institute ( Site 0075), Santa Monica, California
  - University of Colorado Hospital ( Site 0098), Aurora, Colorado
  - Georgetown University Medical Center ( Site 0022), Washington D.C., District of Columbia
  - Emory School of Medicine ( Site 0006), Atlanta, Georgia
  - John H. Stroger Jr. Hospital of Cook County ( Site 1551), Chicago, Illinois
  - University of Chicago ( Site 0068), Chicago, Illinois
  - Parkview Cancer Institute ( Site 0077), Fort Wayne, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center ( Site 0004), Indianapolis, Indiana
  - Wichita Urology Group ( Site 0059), Wichita, Kansas
  - Tulane University School of Medicine ( Site 0088), New Orleans, Louisiana
  - New England Cancer Specialists ( Site 0070), Westbrook, Maine
  - Greater Baltimore Medical Center ( Site 0014), Baltimore, Maryland
  - Dana-Farber Cancer Institute ( Site 1596), Boston, Massachusetts
  - M Health Fairview Ridges Hospital ( Site 1555), Burnsville, Minnesota
  - Morristown Medical Center ( Site 0015), Morristown, New Jersey
  - UNM Comprehensive Cancer Center-Clinical Research Office ( Site 0045), Albuquerque, New Mexico
  - Northwell Health - Monter Cancer Center ( Site 0083), Lake Success, New York
  - New York University Perlmutter Cancer Center ( Site 0008), New York, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0031), New York, New York
  - Cleveland Clinic Main ( Site 1576), Cleveland, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC ( Site 0021), Tulsa, Oklahoma
  - Providence Portland Medical Center [Portland, OR] ( Site 0095), Portland, Oregon
  - MidLantic Urology ( Site 0089), Bala-Cynwyd, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania ( Site 0074), Philadelphia, Pennsylvania
  - Thomas Jefferson University ( Site 1579), Philadelphia, Pennsylvania
  - Fox Chase Cancer Center ( Site 0055), Philadelphia, Pennsylvania
  - Allegheny General Hospital ( Site 0048), Pittsburgh, Pennsylvania
  - Bon Secours St. Francis Health System ( Site 1572), Greenville, South Carolina
  - Carolina Urologic Research Center ( Site 0062), Myrtle Beach, South Carolina
  - Urology Associates [Nashville, TN] ( Site 0053), Nashville, Tennessee
  - Vanderbilt University Medical Center ( Site 0017), Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center ( Site 1552), Dallas, Texas
  - Inova Schar Cancer Institute ( Site 0007), Fairfax, Virginia
  - Charleston Area Medical Center ( Site 0023), Charleston, West Virginia
- Asociación de Beneficencia Hospital Sirio Libanés ( Site 2102), Buenos Aires, Buenos Aires F.D., Argentina
- Australia (6):
  - Western Sydney Local Health District ( Site 1259), Blacktown, New South Wales
  - Macquarie University ( Site 1251), Macquarie Park, New South Wales
  - Cairns Base Hospital ( Site 1257), Cairns, Queensland
  - Mater Misericordiae Ltd ( Site 1258), South Brisbane, Queensland
  - Eastern Health ( Site 1255), Box Hill, Victoria
  - Monash Health ( Site 1260), Clayton, Victoria
- Belgium (6):
  - UCL Saint-Luc - Oncologie Medicale ( Site 0357), Brussels, Bruxelles-Capitale, Region de
  - CHU UCL Namur Site de Godinne ( Site 0354), Yvoir, Namur
  - AZ Maria Middelares Gent ( Site 0353), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 0361), Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge ( Site 0352), Bruges, West-Vlaanderen
  - AZ Delta vzw-Oncology ( Site 0362), Roeselare, West-Vlaanderen
- Canada (11):
  - Arthur J.E. Child Comprehensive Cancer Centre ( Site 0100), Calgary, Alberta
  - BC Cancer Vancouver-Clinical Trials Unit ( Site 0121), Vancouver, British Columbia
  - Silverado Resarch Inc. ( Site 0111), Victoria, British Columbia
  - Moncton Hospital - Horizon Health Network ( Site 0112), Moncton, New Brunswick
  - Sunnybrook Research Institute ( Site 0110), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0107), Toronto, Ontario
  - CIUSSS du Saguenay-Lac-St-Jean ( Site 0116), Chicoutimi, Quebec
  - CIUSSS de l Est de L Ile de Montreal - Hopital Maisonneuve-Rosemont ( Site 0105), Montreal, Quebec
  - Jewish General Hospital ( Site 0120), Montreal, Quebec
  - McGill University Health Centre ( Site 0123), Montreal, Quebec
  - CIUSSS de l'Estrie-CHUS ( Site 0106), Sherbrooke, Quebec
- Colombia (5):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 2003), Medellín, Antioquia
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 2002), Bogotá, Bogota D.C.
  - IMAT S.A.S ( Site 2001), Montería, Departamento de Córdoba
  - Fundación Cardiovascular de Colombia ( Site 2004), Piedecuesta, Santander Department
  - Fundacion Valle del Lili- CIC-Fundacion Valle del Lili ( Site 2005), Cali, Valle del Cauca Department
- Denmark (4):
  - Rigshospitalet University Hospital ( Site 0411), Copenhagen, Capital Region
  - Herlev og Gentofte Hospital. ( Site 0412), Herlev, Capital Region
  - Aarhus University Hospital Skejby ( Site 0418), Aarhus, Central Jutland
  - Odense Universitetshospital ( Site 0413), Odense, Region Syddanmark
- France (16):
  - Hopital de la Timone ( Site 0489), Marseille, Bouches-du-Rhone
  - Centre Georges Francois Leclerc ( Site 0488), Dijon, Bourgogne-Franche-Comté
  - Centre Francois Baclesse ( Site 0459), Caen, Calvados
  - CHU Jean Minjoz ( Site 0455), Besançon, Doubs
  - Institut de Cancerologie du Gard - CHU Caremeau ( Site 0490), Nîmes, Gard
  - CHU de Bordeaux- Hopital Saint Andre ( Site 0456), Bordeaux, Gironde
  - Institut Claudius Regaud IUCT Oncopole ( Site 0486), Toulouse, Haute-Garonne
  - CHU de Montpellier - Hopital Saint-Eloi ( Site 0469), Montpellier, Herault
  - C.H.R.U. de Rennes. Hopital de Pontchaillou ( Site 0492), Rennes, Ille-et-Vilaine
  - CHU Hotel Dieu Nantes ( Site 0458), Nantes, Loire-Atlantique
  - Hopital Belle Isle ( Site 0452), Vantoux, Moselle
  - C.H.U. Lyon Sud ( Site 0466), Pierre-Bénite, Rhone
  - Institut Gustave Roussy ( Site 0487), Villejuif, Val-de-Marne
  - CHU Cochin ( Site 0475), Paris
  - Hopital Europeen Georges Pompidou ( Site 0476), Paris
  - Hopital Bichat du Paris ( Site 0462), Paris
- Germany (11):
  - Klinikum Stuttgart - Katharinenhospital ( Site 0520), Stuttgart, Baden-Wurttemberg
  - Klinikum der Eberhard-Karls-Universitaet Tuebingen ( Site 0549), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen ( Site 0546), Erlangen, Bavaria
  - Klinikum der Universitaet Muenchen - Grosshadern ( Site 0548), Munich, Bavaria
  - Universitaetsklinikum Wuerzburg ( Site 0547), Würzburg, Bavaria
  - Universitaetsklinikum Bonn ( Site 0550), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus ( Site 0532), Dresden, Saxony
  - Universitaetsklinikum Magdeburg A.o.R. ( Site 0535), Magdeburg, Saxony-Anhalt
  - SRH Wald-Klinikum Gera-Zentrum für klinische Studien ( Site 0533), Gera, Thuringia
  - Vivantes Klinikum am Urban ( Site 0529), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf-Onkologisches Zentrum ( Site 0528), Hamburg
- Hungary (5):
  - SZTE Szent-Gyorgyi Albert Klinikai Kozpont ( Site 1010), Szeged, Csongrád megye
  - Bajcsy Zsilinszki Korhaz es Rendelointezet ( Site 1001), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 1006), Debrecen
  - Petz Aladar Megyei Oktato Korhaz ( Site 1012), Győr
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 1007), Kaposvár
- Ireland (2):
  - Tallaght University Hospital ( Site 0734), Dublin
  - University Hospital Waterford ( Site 0747), Waterford
- Israel (10):
  - Ha Emek Medical Center ( Site 0843), Afula
  - Soroka Medical Center ( Site 0849), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0845), Haifa
  - Shaare Zedek Medical Center ( Site 0842), Jerusalem
  - Hadassah Ein Kerem Medical Center ( Site 0841), Jerusalem
  - Meir Medical Center ( Site 0846), Kfar Saba
  - Rabin Medical Center ( Site 0847), Petah Tikva
  - Sheba Medical Center ( Site 0844), Ramat Gan
  - Sourasky Medical Center ( Site 0850), Tel Aviv
  - Yitzhak Shamir Medical Center. ( Site 0848), Ẕerifin
- Italy (10):
  - Policlinico Gemelli di Roma ( Site 0558), Roma, Abruzzo
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga-SCDU Oncologia Medica ( Site 0563), Orbassano, Piedmont
  - AULSS8 Berica-Ospedale S.Bortolo-ONCOLOGIA CLINICA ( Site 0562), Vicenza, Veneto
  - Azienda USL 8 di Arezzo-Medical Oncology ( Site 0565), Arezzo
  - A.O.U. Policlinico Vittorio Emanuele - Presidio Gaspare Rodolico ( Site 0559), Catania
  - Ospedale San Raffaele-Oncologia Medica ( Site 0561), Milan
  - Istituto Nazionale Studio e Cura dei Tumori ( Site 0551), Milan
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori ( Site 0552), Napoli
  - Fondazione Salvatore Maugeri IRCCS ( Site 0554), Pavia
  - Azienda Ospedaliera Santa Maria Terni-S.C. Oncologia Medica e Traslazionale ( Site 0564), Terni
- Japan (18):
  - National Cancer Center Hospital East ( Site 2305), Kashiwa, Chiba
  - University of Tsukuba Hospital ( Site 2302), Tsukuba, Ibaraki
  - St. Marianna University Hospital ( Site 2321), Kawasaki, Kanagawa
  - Kitasato University Hospital ( Site 2306), Sagamihara, Kanagawa
  - Yokosuka Kyosai Hospital ( Site 2307), Yokosuka, Kanagawa
  - Tohoku University Hospital ( Site 2301), Sendai, Miyagi
  - Nagano Municipal Hospital ( Site 2309), Tomitake, Nagano
  - Nara Medical University Hospital ( Site 2312), Kashihara, Nara
  - Osaka Rosai Hospital ( Site 2320), Sakai, Osaka
  - Saitama Prefectural Cancer Center ( Site 2319), Ina-machi, Saitama
  - Dokkyo Medical University Saitama Medical Center ( Site 2304), Koshigaya, Saitama
  - Hamamatsu University Hospital ( Site 2311), Hamamatsu, Shizuoka
  - Institute of Science Tokyo Hospital ( Site 2303), Bunkyō, Tokyo
  - Toranomon Hospital ( Site 2322), Minato-ku, Tokyo
  - Toyama University Hospital ( Site 2308), Toyoma, Toyama
  - Gifu University Hospital ( Site 2310), Gifu
  - Kagoshima University Hospital ( Site 2317), Kagoshima
  - Nagasaki University Hospital ( Site 2315), Nagasaki
- Malaysia (3):
  - University Malaya Medical Centre ( Site 1702), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 1703), George Town, Pulau Pinang
  - Sarawak General Hospital ( Site 1701), Kuching, Sarawak
- Mexico (6):
  - Centro de Urologia Avanzada del Noreste S.A. de C.V. ( Site 0253), Monterrey, Nuevo León
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V. ( Site 0300), Aguascalientes
  - Centro Estatal de Cancerologia de Chihuahua ( Site 0254), Chihuahua City
  - Centro de Tratamiento de Cancer ( Site 0266), Metepec
  - Hospital Angeles Roma ( Site 0262), Mexico City
  - Instituto Nacional de Cancerologia. ( Site 0256), Mexico City
- Philippines (3):
  - THE MEDICAL CITY ILOILO ( Site 1756), Iloilo City, Iloilo
  - The Medical City ( Site 1752), Pasig, National Capital Region
  - St. Luke s Medical Center ( Site 1751), Quezon City, National Capital Region
- Poland (9):
  - Clinical Research Center Medic-R ( Site 1073), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im.prof. F. Lukaszczyka w Bydgoszczy ( Site 1068), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Szpital Wojewodzki ( Site 1062), Tarnów, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego ( Site 1063), Wroclaw, Lower Silesian Voivodeship
  - Europejskie Centrum Zdrowia Otwock ( Site 1058), Otwock, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 1051), Warsaw, Masovian Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1072), Bialystok, Podlaskie Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku ( Site 1057), Słupsk, Pomeranian Voivodeship
  - Beskidzkie Centrum Onkologii im. Jana Pawla II ( Site 1061), Bielsko-Biala, Silesian Voivodeship
- Russia (17):
  - Clinic of Bashkortostan State Medical University ( Site 0873), Ufa, Baskortostan, Respublika
  - Ivanovo Regional Oncology Dispensary ( Site 0852), Ivanovo, Ivanovo Oblast
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0861), Krasnoyarsk, Krasnoyarsk Krai
  - Kursk Regional Clinical Oncology Dispensary ( Site 0854), Kursk, Kursk Oblast
  - Russian Oncological Research Center n.a. N.N.Blokhin of MoH ( Site 0878), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 0884), Moscow, Moscow
  - Central Clinical Hospital with outpatient Clinic ( Site 0856), Moscow, Moscow
  - Bayandin Murmansk Regional Clinical Hospital ( Site 0859), Murmansk, Murmansk Oblast
  - Volga District Medical Center Federal Medical and Biological Agency ( Site 0857), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Omsk Clinical Oncology Dispensary ( Site 0865), Omsk, Omsk Oblast
  - Leningrad Regional Oncology Center ( Site 0868), Saint Petersburg, Sankt-Peterburg
  - Clinical Hospital Saint Luka ( Site 0867), Saint Petersburg, Sankt-Peterburg
  - First St. Petersburg State Medical University n.a. acad. I.P. Pavlov ( Site 0872), Saint Petersburg, Sankt-Peterburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 0860), Saint Petersburg, Sankt-Peterburg
  - Saratov State Medical University n.a. V.I.Razumovskiy ( Site 0866), Saratov, Saratov Oblast
  - Sverdlovsk Regional Oncology Hospital ( Site 0874), Yekaterinburg, Sverdlovsk Oblast
  - Medical Sanitary Unit Neftyannik ( Site 0888), Tyumen, Tyumen Oblast
- Singapore (2):
  - National University Hospital ( Site 1802), Singapore, Central Singapore
  - Tan Tock Seng Hospital ( Site 1804), Singapore, Central Singapore
- South Africa (2):
  - Steve Biko Academic Hospital-Medical Oncology ( Site 1601), Pretoria, Gauteng
  - Groote Schuur Hospital ( Site 1602), Cape Town, Western Cape
- South Korea (7):
  - National Cancer Center ( Site 1354), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 1356), Seongnam-si, Kyonggi-do
  - Asan Medical Center ( Site 1355), Songpagu, Seoul
  - Kyungpook National University Chilgok Hospital-Urology ( Site 1357), Deagu, Taegu-Kwangyokshi
  - Korea University Anam Hospital ( Site 1351), Seoul
  - Seoul National University Hospital ( Site 1352), Seoul
  - Samsung Medical Center ( Site 1353), Seoul
- Spain (11):
  - Hosp. Gral. Universitari Germans Trias i Pujol ( Site 0675), Badalona, Barcelona
  - Hospital Clinic i Provincial ( Site 0674), Barcelona, Catalonia
  - Hospital San Pedro de Alcantara ( Site 0697), Cáceres, Extremadura
  - Institut Català d'Oncologia (ICO) - Girona ( Site 0700), Girona, Gerona
  - Hospital Universitario Quiron Madrid ( Site 0694), Pozuelo de Alarcón, Madrid, Comunidad de
  - Instituto Valenciano de Oncologia - IVO ( Site 0679), Valencia, Valenciana, Comunitat
  - Hospital del Mar ( Site 0698), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 0691), Madrid
  - Hospital Universitario San Carlos ( Site 0678), Madrid
  - Hospital Universitario la Paz ( Site 0690), Madrid
  - Hospital de Nuestra Senora de Valme ( Site 0693), Seville
- Sweden (5):
  - Laenssjukhuset Ryhov ( Site 1215), Jönköping, Jönköping County
  - Karolinska Universitetssjukhuset Solna ( Site 1212), Stockholm, Stockholm County
  - Akademiska Sjukhuset ( Site 1211), Uppsala, Uppsala County
  - Cancercentrum ( Site 1214), Umeå, Västerbotten County
  - Onkologiska kliniken ( Site 1217), Gothenburg, Västra Götaland County
- Thailand (4):
  - Ramathibodi Hospital. ( Site 1451), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 1452), Bangkok, Bangkok
  - Maharaj Nakorn Chiangmai Hospital ( Site 1453), Chiang Mai
  - Srinagarind Hospital ( Site 1454), Khon Kaen
- Turkey (Türkiye) (7):
  - Hacettepe Universitesi Tıp Fakultesi ( Site 0931), Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0930), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 0926), Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi ( Site 0921), Istanbul
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi ( Site 0929), Konya
  - Sakarya Universitesi Tip Fakultesi ( Site 0933), Sakarya
  - Karadeniz Teknik Universitesi Tip Fakultesi Farabi Hastanesi ( Site 0924), Trabzon
- Ukraine (12):
  - Cherkasy Regional Oncology Dispensary ( Site 0959), Cherkasy, Cherkasy Oblast
  - MNPE City Clinical Hospital #4 of Dnipro Regional Council ( Site 0951), Dnipro, Dnipropetrovsk Oblast
  - ME І.І. Mechnykov Dnipro Regional Clinical Hospital ( Site 0963), Dnipropetrovsk, Dnipropetrovsk Oblast
  - Regional Oncology Center of Kharkiv ( Site 0958), Kharkiv, Kharkivs’ka Oblast’
  - MNPE V.I. Shapoval Regional Medical Clinical Urology and Nephrology Center of KharkivRegCouncil ( Site 0969), Kharkiv, Kharkivs’ka Oblast’
  - Municipal Non-profit Enterprise of Kharkiv Regional Council RCSDRPP ( Site 0973), Kharkiv, Kharkivs’ka Oblast’
  - Communal nonprofit enterprise "Kherson Regional Oncology Dispensary" of Kherson Regional Council ( Site 0976), Antonivka Village, Kherson Oblast
  - SNPE National Cancer Institute ( Site 0962), Kyiv, Kyivska Oblast
  - MNPE Lviv Regional Clinical Hospital of Lviv Regional Council ( Site 0955), Lviv, Lviv Oblast
  - Lviv State Regional Oncological Center ( Site 0967), Lviv, Lviv Oblast
  - Zhytomyr Regional Oncology Center ( Site 0971), Zhytomyr, Zhytomyr Oblast
  - Kyiv City Clinical Oncology Center ( Site 0960), Kyiv
- United Kingdom (10):
  - Walsall Manor Hospital-Oncology ( Site 0743), Walsall, Devon
  - Kent and Canterbury Hospital ( Site 0733), Canterbury, England
  - The James Cook University Hospital ( Site 0730), Middlesbrough, England
  - Imperial College Healthcare NHS Trust ( Site 0745), London, Hammersmith and Fulham
  - Lister Hospital ( Site 0739), Stevenage, Hertfordshire
  - Barts Health NHS Trust - St Bartholomew s Hospital ( Site 0725), London, London, City of
  - The Royal Marsden Foundation Trust ( Site 0726), London, London, City of
  - Western General Hospital ( Site 0749), Edinburgh, Midlothian
  - Clatterbridge Oncology Centre ( Site 0731), Metropolitan Borough of Wirral
  - Royal Cornwall Hospital ( Site 0727), Truro

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Galsky MD, Hoimes CJ, Necchi A, Shore N, Witjes JA, Steinberg G, Bedke J, Nishiyama H, Fang X, Kataria R, Sbar E, Jia X, Siefker-Radtke A. Perioperative pembrolizumab therapy in muscle-invasive bladder cancer: Phase III KEYNOTE-866 and KEYNOTE-905/EV-303. Future Oncol. 2021 Aug;17(24):3137-3150. doi: 10.2217/fon-2021-0273. Epub 2021 May 19. PMID 34008425
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26129&tenant=MT_MSD_9011